CLINICAL TRIAL: NCT05385367
Title: Life Cycle Assessment of General Anesthetic, Regional Anesthetic and the Combination of General Anesthetic and Regional Anesthetic: a Randomized Controlled Trial
Brief Title: Life Cycle Assessment of Different Types of Anesthetic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00118522
Record Dates: First submitted 2022-05-11; First posted 2022-05-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Carbon Footprint in Anesthetic
Keywords: carbon footprint; anesthetic waste; life cycle analsis
MeSH Terms: interventions — Anesthetics, General

STUDY DESIGN:
Intervention Model Description: Mulicentre trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regional anesthetic (Other): Patients only have nerve block with or without sedation
  Interventions: Other: Regional anesthetic
- General anesthetic (Other): Patients only have general anesthetic
  Interventions: Other: General anesthetic
- Combined general anesthetic and regional anesthetic (Other): Patients have both general anesthetic and regional anesthetic together
  Interventions: Other: Combined general anesthetic and regional anesthetic

INTERVENTIONS:
Other: Regional anesthetic — Patient having just the nerve block for surgery
  Arms: Regional anesthetic
Other: General anesthetic — Patient having just general anesthetic ie. 'go completely under' for surgery
  Arms: General anesthetic
Other: Combined general anesthetic and regional anesthetic — Patient having a combination of a nerve block and general anesthetic for surgery
  Arms: Combined general anesthetic and regional anesthetic

SUMMARY:
Following Ethics approval, all adult patients undergoing surgery to fix the wrist fracture will be approached and consent to undergo this study. The amount of waste generated from general anesthetic, regional anesthetic and regional+general anesthetic will be collected and weighed.

Patients undergoing this type of wrist surgery have only regional anesthetic, or general anesthetic, or both ie. regional anesthetic and general anesthetic.

The aim of the study is to compare the amount of waste generated from each type of anesthetic and this will give us a better idea of which anesthetic is more environmentally sustainable.

DETAILED DESCRIPTION:
Following Ethics approval, all adult patients undergoing surgery to fix the wrist fracture will be approached and consent to undergo this study. The amount of waste generated from general anesthetic, regional anesthetic and regional+general anesthetic will be collected and weighed. Waste will include disposable and reusable wastes. Examples of disposable waste are all plastic packaging, syringes, needles, breathing tube, breathing circuits, gloves as well as drugs. Examples of reusable waste will be anesthetic face mask, laryngeal mask (which is a form of airway device that can be reprocessed), sterile gowns. The amount of anesthetic gas used will be obtained from the anesthetic machine.

Patients undergoing this type of wrist surgery have only regional anesthetic (freezing performed higher up in the arm to numb the whole arm for several hours), or general anesthetic (patient completely goes to deep anesthetic sleep), or both ie. regional anesthetic (freezing just for pain control afterwards) and general anesthetic (patient goes to deep anesthetic sleep after the freezing is done and they may need less pain killer during the surgery as well as afterwards).

The amount of waste generated will be compared amongst these 3 groups by life cycle analysis.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing open reduction and internal fixation of wrist
* ASA 1-3

Exclusion Criteria:

* no contraindications for general anesthetic in the group for general anesthetic and vice versa

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Carbon dioxide emission | During surgical intervention
  Amount of carbon dioxide emission

SECONDARY OUTCOMES:
Generation of solid waste | During surgical intervention
  Solid waste generated within the type of anesthetic
Duration of surgery | During surgical intervention
  Duration of surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta